CLINICAL TRIAL: NCT00013013
Title: A Randomized Trial to Implement the AHCPR Smoking Cessation Guideline
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CPG 97-039
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Smoking; Smoking Cessation
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Procedure: Systems Support

INTERVENTIONS:
Procedure: Systems Support

SUMMARY:
Among veterans, smoking is the single most important risk factor for preventable mortality and morbidity, and studies suggest a higher prevalence of smoking among veterans than the general population. The VHA has encouraged adoption of the AHCPR Guideline for Smoking Cessation, yet most hospitals have poorly developed smoking cessation programs.

DETAILED DESCRIPTION:
Background:

Among veterans, smoking is the single most important risk factor for preventable mortality and morbidity, and studies suggest a higher prevalence of smoking among veterans than the general population. The VHA has encouraged adoption of the AHCPR Guideline for Smoking Cessation, yet most hospitals have poorly developed smoking cessation programs.

Objectives:

The present study is designed to investigate the effectiveness of an organizational strategy to increase compliance with the AHCPR guideline. Short term goals of the study include increasing the rate of identification of smokers and increasing the delivery of brief smoking cessation interventions. Long term goals include reducing tobacco consumption among veterans.

Methods:

Twenty VAMC�s with active primary care clinics have been randomly assigned to either control (usual practice; UP) or intervention (organizational support; OS) groups. The intervention hospitals receive staff training and site consultation; all hospitals will receive the AHCPR guideline. Rate of identification of smokers in the medical record, smoking cessation rates, provision of smoking cessation services (e.g., NRT, counseling), and costs of NRT will be determined via telephone interviews with patients, chart review, and electronic records.

Status:

Baseline data collection is nearly complete, and the intervention period will be complete in September, 2000. We have completed telephone surveys with approximately 4500 veterans. Analysis of study data is ongoing, and manuscript preparation will begin within the next few months.

ELIGIBILITY:
Inclusion Criteria:

Subjects must be smokers.

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Study Completion 2001-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne M. Joseph, MD MPH, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Joseph AM, Arikian NJ, An LC, Nugent SM, Sloan RJ, Pieper CF; GIFT Research Group. Results of a randomized controlled trial of intervention to implement smoking guidelines in Veterans Affairs medical centers: increased use of medications without cessation benefit. Med Care. 2004 Nov;42(11):1100-10. doi: 10.1097/00005650-200411000-00009. PMID 15586837